CLINICAL TRIAL: NCT01117311
Title: The Effect of Vagal Nerve Stimulation on Enteroendocrine Secretion and Glucose Metabolism
Brief Title: Vagal Nerve Stimulation and Glucose Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Principal Investigator, Adrian Vella, Professor of Medicine, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 09-008825; R01DK082396 (NIH); UL1RR024150 (NIH)
Record Dates: First submitted 2010-05-04; First posted 2010-05-05 (Estimated); Results first posted 2014-01-06 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2013-11

CONDITIONS: Type 2 Diabetes; Obesity; Gastric Emptying
Keywords: Vagus; Diabetes; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- VNB off first, then VNB on (Experimental): Subjects assigned to this reporting group had the vagal nerve blocker (VNB) on for the lead in period (Mixed Meal 1), then VNB off first for the first intervention (Mixed Meal 2), then VNB on for the second intervention (Mixed Meal 3).
  Interventions: Device: VNB on; Device: VNB off
- VNB on first, then VNB off (Experimental): Subjects assigned to this reporting group had the vagal nerve blocker (VNB) on for the lead in period (Mixed Meal 1), then VNB on first for the first intervention (Mixed Meal 2), then VNB off for the second intervention (Mixed Meal 3).
  Interventions: Device: VNB on; Device: VNB off

INTERVENTIONS:
Device: VNB on — The implanted Vagal Nerve Blocker will be on at the time of study.
Device: VNB off — The implanted Vagal Nerve Blocker will be off at the time of study.

SUMMARY:
The overall aim of this application is to determine the mechanism(s) by which common bariatric surgical procedures alter carbohydrate metabolism. The study proposed will examine the effect of vagal nerve stimulation on insulin secretion and action.

DETAILED DESCRIPTION:
The overall aim of this application is to determine the mechanism(s) by which common bariatric surgical procedures alter carbohydrate metabolism. Very often, resolution of diabetes occurs in the early post-operative period prior to the development of significant weight loss. It has been suggested that bariatric surgery alters insulin action but few studies have examined insulin secretion or postprandial glucose fluxes in such patients. At the present time, little is known about how the various bariatric surgical procedures alter glucose homeostasis. It is essential that the effect of bariatric surgery and meal size on these parameters be understood and accurately measured. Enteroendocrine secretion is affected by the rate of intestinal delivery of calories and may also be modulated by the enteric nervous system and the rate of direct delivery of nutrients to enteroendocrine cells. Direct measurement of intestinal transit is also an important part of understanding how bariatric surgery alters intestinal secretion of hormones that may alter glucose metabolism. The Oral and C-peptide Minimal Models when applied to C-peptide, glucose and insulin concentrations after ingestion of a standard labeled mixed meal can accurately measure insulin secretion and action. Subsequently, the disposition index provides a measurement of the appropriateness of insulin secretion for the prevailing insulin action. When coupled with established triple-tracer methodology, a mixed meal can be used to measure fasting and postprandial glucose fluxes. Though the vagal trunks are preserved during bariatric surgery, gastric transection during the formation of a gastric pouch for Roux-en-Y gastric bypass (RYGB), or during the sleeve gastrectomy for the duodenal switch procedure, may denervate post-gastric organs including the pancreas and intestine. Reversible vagal block results in weight loss, decreased caloric intake, earlier satiation and reduced hunger. The effect of this form of vagal denervation on glycemic control is unclear. There is evidence that hepatic parasympathetic input regulates insulin action in rodents. Vagal afferents are also important in hepatoportal glucose sensing.

Subjects enrolled into the study would be on stable Vagal Nerve Stimulation Blocker (VNB) intervention in excess of 12 months, having taken part in prior observational study examining the long-term effects of vagal inhibition. All subjects will be studied three times after using a mixed meal. Participants will be admitted to the Mayo Clinic Clinical Research Unit at 17.00 hours the evening before the study. Following ingestion of a standardized low calorie mixed meal (400 Kcal: 55% carbohydrate, 30% fat, and 15% protein) subjects will fast overnight. During the experiment subjects will undergo a mixed meal study as outlined below (Lead-in Mixed Meal 1). On the day after study, subjects will be randomized to one of 2 interventions: either discontinue use of the VNB or continue its use. Subjects will then be restudied (Mixed Meal 2) the day after admission to the Clinical Research Unit at 17.00 hours on the 13th day after randomization. To determine the metabolic effects, if any, of starting VNB therapy, on the day after study, VNB use will be resumed or discontinued depending on prior activation or inactivation. Subjects will then be restudied (Mixed Meal 3) the day after admission to the Clinical Research Unit at 17.00 hours on the 13th day after completion of Mixed Meal 2. Following completion of the study, VNB use will be resumed in all subjects.

ELIGIBILITY:
Previous Implantation of a Vagal Nerve Stimulator for obesity as part of a prior study examining the effect of vagal nerve stimulator on obesity

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2011-03; Primary Completion 2012-06 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Vella, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects will be recruited out of the study population for a previous multi-center observational study examining the long-term effects of vagal stimulation. In this previous study the Vagal Nerve Blocker (VNB) was implanted.
Pre-assignment Details: 9 subjects were screened and enrolled, but 2 subjects did not return after the screening visit.
Groups:
- VNB Off First, Then VNB on: Subjects assigned to this reporting group had the vagal nerve blocker (VNB) off first for the first intervention (Mixed Meal 2), then VNB on for the second intervention (Mixed Meal 3).
- VNB on First, Then VNB Off: Subjects assigned to this reporting group had the vagal nerve blocker (VNB) on first for the first intervention (Mixed Meal 2), then VNB off for the second intervention (Mixed Meal 3).
Period: Lead-in Mixed Meal 1
Arm/Group | VNB Off First, Then VNB on | VNB on First, Then VNB Off
Started | 3 | 4
Completed | 3 | 4
Not Completed | 0 | 0
Period: First Intervention - Mixed Meal 2
Arm/Group | VNB Off First, Then VNB on | VNB on First, Then VNB Off
Started | 3 | 4
Completed | 3 | 4
Not Completed | 0 | 0
Period: Second Intervention - Mixed Meal 3
Arm/Group | VNB Off First, Then VNB on | VNB on First, Then VNB Off
Started | 3 | 4
Completed | 3 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes groups randomized to have the VNB off first and the VNB on first.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 53.1 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Disposition Index
Description: Total Disposition Index (DI) is a calculated value which represents the ability of a person's pancreas to lower blood glucose. A higher number means the pancreas is better able to lower blood glucose and a lower number means the pancreas is less able to lower blood glucose.
Time Frame: baseline, 2 weeks
Measure: Mean (Standard Error); unit: 10^-14dl/kg/min^2 per pmol/l
Arm/Group | VNB on | VNB Off
Number analyzed (Participants) | 7 | 7
10^-14dl/kg/min^2 per pmol/l | 703 (240) | 532 (145)

2. Secondary Outcome: Gastric Emptying Half-time
Description: Gastric emptying half time is the time for half of the ingested solids or liquids to leave the stomach.
Time Frame: approximately 2 hours after radiolabeled meal is ingested
Measure: Mean (Standard Error); unit: minutes
Arm/Group | VNB on | VNB Off
Number analyzed (Participants) | 7 | 7
minutes | 167 (17) | 160 (23)

ADVERSE EVENTS:
Arm/Group | VNB Off | VNB on
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/7 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No